CLINICAL TRIAL: NCT05559463
Title: Effect of Anti-inflammatory (ITIS) Diet in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Monica Guma, Associate Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161474_2
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ITIS diet (Experimental): anti-inflammatory (ITIS) diet for 28 days
  Interventions: Dietary Supplement: ITIS diet

INTERVENTIONS:
Dietary Supplement: ITIS diet — anti-inflammatory (ITIS) diet for 28 days

SUMMARY:
To study the effect of anti-inflammatory diet on clinical and biological outcomes in patients with knee osteoarthritis

DETAILED DESCRIPTION:
The investigators would like to evaluate how inflammation occurs in the joints of subjects with osteoarthritis, and identify molecules and bacteria that can predict whether a patients with knee osteoarthritis will have more or less pain . Blood, urine and stool will be evaluated in the laboratory and compared to their own samples after changes in diet. This is an exploratory study, which is meant to gather preliminary data about the quick effects of changes in diet and treatment on molecules in blood/urine and bacteria in stools. These studies can provide clues to the cause of disease and might ultimately lead to new therapies.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed of Knee Ostoeaarthritis
* without changes in treatment in the last 3 months

Exclusion Criteria:

* food allergies
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of baseline pain measured by visual analogue scale (0-10) after 28 days | 28 days
  Change of baseline pain measured by visual analogue scale (0-10) after 28 days, being 0 no pain, and 10 the worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sala-Climent M, Bu K, Coras R, Cedeno M, Zuffa S, Murillo-Saich J, Mannochio-Russo H, Allaband C, Hose MK, Quan A, Choi SI, Nguyen K, Golshan S, Blank RB, Holt T, Lane NE, Knight R, Scher J, Dorrestein P, Clemente J, Guma M. Targeted Microbial Shifts and Metabolite Profiles Were Associated with Clinical Response to an Anti-Inflammatory Diet in Osteoarthritis. Nutrients. 2025 Aug 22;17(17):2729. doi: 10.3390/nu17172729. PMID 40944120